CLINICAL TRIAL: NCT03893500
Title: Utility of Device and App-based Mobile Health Monitoring as a Tool for Evaluation of Clinical Response to Therapies in Pulmonary Arterial Hypertension
Brief Title: Utility of At-home Monitoring of Exercise Capacity by App-based 6-minute Walk Test
Acronym: DynAMITE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: PHaware (Unknown)
Responsible Party: Principal Investigator, Roham T. Zamanian, Associate Professor of Medicine, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-DynAMITE; IRB-48742 (Other: Administrative Panel on Human Subjects in Medical Research)
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Six minute walk test; Six minute walk distance; Heart rate recovery; Mobile health
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Initiating a new PAH medication (Experimental): Participants will start a new PAH medication
  Interventions: Device: Home-based 6 minute walk test
- Continuing previous PAH medication regimen (Active Comparator): Participants will continue the medication regimen that they were on prior to enrollment
  Interventions: Device: Home-based 6 minute walk test

INTERVENTIONS:
Device: Home-based 6 minute walk test — Participants will receive a loaner Apple Watch with the Walk.Talk.Track. (WTT, produced by PHaware) app downloaded. Participants will perform a daily 6MWT at home using the Apple Watch and WTT app. They will undergo a history and physical, blood draw, echocardiogram and in-clinic 6MWT at the baseline and 12-week follow up visit.

SUMMARY:
* Evaluate for accuracy and reproducibility of data collected via the participant-operated Walk.Talk.Track. (WTT) app combined with Apple Watch during in-clinic, technician proctored 6MWT's.

  * Determine whether the WTT app on the Apple Watch can accurately collect information on distance traveled and heart rate (HR) during in-clinic 6MWT run by American Thoracic Society (ATS) guidelines
  * Determine whether participants can operate the WTT app and Apple Watch effectively to gather accurate data in a monitored and home-based setting
* Prospectively monitor for changes in WTT app recorded 6MWT results following initiation of therapy in a treatment naïve cohort of PAH participants

  * Evaluate whether changes from baseline in 6 minute walk distance (6MWD) and heart rate recovery at one minute (HRR1) as well as other variables that have been associated with disease severity in PAH and left-sided heart disease (resting HR, heart rate variability [HRV], chronotropic index [CI]) can be identified before the 12-week follow up when comparing the treatment arm and the control arm
  * Evaluate whether changes from baseline in the HRR1, resting HR, HRV and/or CI are more evident in treatment responders when compared to treatment non-responders.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of WHO Group I Pulmonary Arterial Hypertension (PAH) (Idiopathic (I)PAH, Heritable PAH (including Hereditary Hemorrhagic Telangiectasia), Associated (A)PAH (including collagen vascular disorders, drugs+toxins exposure, congenital heart disease, and portopulmonary disease).
* Do not meet exclusion criteria

Exclusion Criteria:

* Pulmonary Hypertension due to left heart disease (PH-LHD, WHO group 2), Pulmonary hypertension due to chronic lung disease (PH-CLD, WHO group 3), Chronic thrombo-embolic pulmonary hypertension (CTEPH, WHO group 4), pulmonary hypertension with unclear and/or multi-factorial mechanisms (WHO goup 5)
* Inability to perform a 6 minute walk test (6MWT)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
App/watch recorded and in-clinic recorded six minute walk distance (6MWD) | 12 weeks
  App/watch recorded and in-clinic recorded 6MWD will be compared by Bland Altman graph and will be considered interchangeable if the line of equality lands within the 95% confidence interval of the mean difference
Count of participants with an increase of >32 meters in 6MWD from baseline as a measure of time to response to therapy | 12 weeks
  Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Count of participants with an increase of >3bpm in heart rate recovery at one minute (HRR1) from baseline as a measure of time to response to therapy | 12 weeks
  HRR1 is calculated as peak heart rate (pHR) - HR one minute into recovery period. Hazard ratios will be calculated at two week intervals to evaluate for between group differences

SECONDARY OUTCOMES:
Count of participants with a decrease of >5bpm in resting HR from baseline as a measure of time to response to therapy | 12 weeks
  Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Count of participants with an increase of >5ms in heart rate variability (HRV) from baseline as a measure of time to response to therapy | 12 weeks
  HRV will be calculated as the standard deviation of R wave to R wave intervals (SDNN) over the 2 minute period following exercise. Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Count of participants with an increase of >5% in chronotropic index (CI) from baseline as a measure of time to response to therapy | 12 weeks
  CI will be calculated as (actual peak HR - resting HR)/(Age predicted peak HR [220-age] - resting HR). Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Within the treatment arm, count of participants with an increase of >3bpm in heart rate recovery at one minute (HRR1) from baseline when comparing medication responders vs non-responders | 12 weeks
  Medication responders will have a ≥32m improvement in 6MWD at 12 weeks; non-responders will have <32m improvement. Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Within the treatment arm, count of participants with a decrease of >5bpm in resting HR from baseline when comparing medication responders vs non-responders | 12 weeks
  Medication responders will have a ≥32m improvement in 6MWD at 12 weeks; non-responders will have <32m improvement. Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Within the treatment arm, count of participants with an increase of >5ms in heart rate variability (HRV) from baseline when comparing medication responders vs non-responders | 12 weeks
  Medication responders will have a ≥32m improvement in 6MWD at 12 weeks; non-responders will have <32m improvement. Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Within the treatment arm, count of participants with an increase of >5% in chronotropic index (CI) from baseline when comparing medication responders vs non-responders | 12 weeks
  Medication responders will have a ≥32m improvement in 6MWD at 12 weeks; non-responders will have <32m improvement. Hazard ratios will be calculated at two week intervals to evaluate for between group differences
Between group difference in 6MWD as a measure of response to the intervention | 12 weeks
  A two-sample T-test will be performed on the delta change in 6MWD (week 12 - baseline / baseline) x100]) between the treatment and control groups and a p-value will be calculated from this data.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoeper MM, Kramer T, Pan Z, Eichstaedt CA, Spiesshoefer J, Benjamin N, Olsson KM, Meyer K, Vizza CD, Vonk-Noordegraaf A, Distler O, Opitz C, Gibbs JSR, Delcroix M, Ghofrani HA, Huscher D, Pittrow D, Rosenkranz S, Grunig E. Mortality in pulmonary arterial hypertension: prediction by the 2015 European pulmonary hypertension guidelines risk stratification model. Eur Respir J. 2017 Aug 3;50(2):1700740. doi: 10.1183/13993003.00740-2017. Print 2017 Aug. PMID 28775047
- [Background] Weatherald J, Boucly A, Sahay S, Humbert M, Sitbon O. The Low-Risk Profile in Pulmonary Arterial Hypertension. Time for a Paradigm Shift to Goal-oriented Clinical Trial Endpoints? Am J Respir Crit Care Med. 2018 Apr 1;197(7):860-868. doi: 10.1164/rccm.201709-1840PP. No abstract available. PMID 29256625
- [Background] Wallen MP, Gomersall SR, Keating SE, Wisloff U, Coombes JS. Accuracy of Heart Rate Watches: Implications for Weight Management. PLoS One. 2016 May 27;11(5):e0154420. doi: 10.1371/journal.pone.0154420. eCollection 2016. PMID 27232714
- [Background] Nogic J, Thein PM, Cameron J, Mirzaee S, Ihdayhid A, Nasis A. The utility of personal activity trackers (Fitbit Charge 2) on exercise capacity in patients post acute coronary syndrome [UP-STEP ACS Trial]: a randomised controlled trial protocol. BMC Cardiovasc Disord. 2017 Dec 29;17(1):303. doi: 10.1186/s12872-017-0726-8. PMID 29284402
- [Background] Zoller D, Siaplaouras J, Apitz A, Bride P, Kaestner M, Latus H, Schranz D, Apitz C. Home Exercise Training in Children and Adolescents with Pulmonary Arterial Hypertension: A Pilot Study. Pediatr Cardiol. 2017 Jan;38(1):191-198. doi: 10.1007/s00246-016-1501-9. Epub 2016 Nov 14. PMID 27841007
- [Background] Cole CR, Blackstone EH, Pashkow FJ, Snader CE, Lauer MS. Heart-rate recovery immediately after exercise as a predictor of mortality. N Engl J Med. 1999 Oct 28;341(18):1351-7. doi: 10.1056/NEJM199910283411804. PMID 10536127
- [Background] Tonelli AR, Wang XF, Alkukhun L, Zhang Q, Dweik RA, Minai OA. Heart rate slopes during 6-min walk test in pulmonary arterial hypertension, other lung diseases, and healthy controls. Physiol Rep. 2014 Jun 11;2(6):e12038. doi: 10.14814/phy2.12038. Print 2014 Jun 1. PMID 24920122
- [Background] Swigris JJ, Olson AL, Shlobin OA, Ahmad S, Brown KK, Nathan SD. Heart rate recovery after six-minute walk test predicts pulmonary hypertension in patients with idiopathic pulmonary fibrosis. Respirology. 2011 Apr;16(3):439-45. doi: 10.1111/j.1440-1843.2010.01877.x. PMID 20946337
- [Background] Ramos RP, Arakaki JS, Barbosa P, Treptow E, Valois FM, Ferreira EV, Nery LE, Neder JA. Heart rate recovery in pulmonary arterial hypertension: relationship with exercise capacity and prognosis. Am Heart J. 2012 Apr;163(4):580-8. doi: 10.1016/j.ahj.2012.01.023. Epub 2012 Mar 30. PMID 22520523
- [Background] Dobre D, Zannad F, Keteyian SJ, Stevens SR, Rossignol P, Kitzman DW, Landzberg J, Howlett J, Kraus WE, Ellis SJ. Association between resting heart rate, chronotropic index, and long-term outcomes in patients with heart failure receiving beta-blocker therapy: data from the HF-ACTION trial. Eur Heart J. 2013 Aug;34(29):2271-80. doi: 10.1093/eurheartj/ehs433. Epub 2013 Jan 12. PMID 23315907
- [Background] Huang RY, Dung LR. Measurement of heart rate variability using off-the-shelf smart phones. Biomed Eng Online. 2016 Jan 29;15:11. doi: 10.1186/s12938-016-0127-8. PMID 26822804
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Latus H, Bandorski D, Rink F, Tiede H, Siaplaouras J, Ghofrani A, Seeger W, Schranz D, Apitz C. Heart Rate Variability is Related to Disease Severity in Children and Young Adults with Pulmonary Hypertension. Front Pediatr. 2015 Jul 7;3:63. doi: 10.3389/fped.2015.00063. eCollection 2015. PMID 26217650
- [Background] Azarbal B, Hayes SW, Lewin HC, Hachamovitch R, Cohen I, Berman DS. The incremental prognostic value of percentage of heart rate reserve achieved over myocardial perfusion single-photon emission computed tomography in the prediction of cardiac death and all-cause mortality: superiority over 85% of maximal age-predicted heart rate. J Am Coll Cardiol. 2004 Jul 21;44(2):423-30. doi: 10.1016/j.jacc.2004.02.060. PMID 15261942
- [Background] Provencher S, Chemla D, Herve P, Sitbon O, Humbert M, Simonneau G. Heart rate responses during the 6-minute walk test in pulmonary arterial hypertension. Eur Respir J. 2006 Jan;27(1):114-20. doi: 10.1183/09031936.06.00042705. PMID 16387943
- [Background] Girotra S, Kitzman DW, Kop WJ, Stein PK, Gottdiener JS, Mukamal KJ. Heart rate response to a timed walk and cardiovascular outcomes in older adults: the cardiovascular health study. Cardiology. 2012;122(2):69-75. doi: 10.1159/000338736. Epub 2012 Jun 20. PMID 22722364
- [Background] Lauer MS, Francis GS, Okin PM, Pashkow FJ, Snader CE, Marwick TH. Impaired chronotropic response to exercise stress testing as a predictor of mortality. JAMA. 1999 Feb 10;281(6):524-9. doi: 10.1001/jama.281.6.524. PMID 10022108
- See also: ATS guidelines for the 6 minute walk test — http://www.thoracic.org/statements/resources/pfet/sixminute.pdf